CLINICAL TRIAL: NCT00316953
Title: A Phase I Study of BMS-354825 (Dasatinib) in Children With Recurrent/Refractory Solid Tumors or Imatinib Resistant Ph+ Leukemia (BMS Trial CA180038)
Brief Title: Dasatinib in Treating Young Patients With Recurrent or Refractory Solid Tumors or Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia or Chronic Myelogenous Leukemia That Did Not Respond to Imatinib Mesylate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01824; ADVL0516; U10CA97452 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000467233 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Childhood Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Meningeal Chronic Myelogenous Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Relapsing Chronic Myelogenous Leukemia; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

ARMS (2):
- Stratum 1 (solid tumors) (Experimental): Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib; Other: pharmacological study; Other: laboratory biomarker analysis
- Stratum 2 (leukemia) (Experimental): Patients receive dasatinib as in stratum 1. Cohorts of 3-12 patients receive escalating or de-escalating doses of dasatinib. The MTD is defined as the dose preceding that at which 7 of 12 patients experience DLT.
  Interventions: Drug: dasatinib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dasatinib — Given orally
  Other Names: BMS-354825; Sprycel
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of dasatinib in treating young patients with recurrent or refractory solid tumors or Philadelphia chromosome-positive acute lymphoblastic leukemia or chronic myelogenous leukemia that did not respond to imatinib mesylate. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicities and estimate the maximum tolerated dose or the recommended phase 2 dose of dasatinib in pediatric patients with refractory solid tumors.

II. Determine the toxicities of dasatinib in pediatric patients with imatinib mesylate-resistant Philadelphia chromosome-positive (Ph+) leukemia.

III. Characterize the pharmacokinetics of dasatinib in pediatric patients with refractory solid tumors or imatinib-resistant Ph+ leukemia.

SECONDARY OBJECTIVES:

I. Preliminarily define the antitumor activity of dasatinib in pediatric patients with refractory solid tumors within the confines of a phase I study.

II. Obtain pilot data on the activity of dasatinib administered in pediatric patients with Ph+ leukemia.

III. Assess the biologic activity of dasatinib on tumor cells when available. IV. Determine the phosphotyrosine state of SRC and ABL substrates and correlate this with dasatinib dosage and antitumor activity (pharmacodynamics study).

OUTLINE: This is a multicenter, dose-escalation study. Patients are stratified according to disease (solid tumors vs leukemia).

Stratum 1 (solid tumors): Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of dasatinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which ≥ 2 of 6 patients experience dose-limiting toxicity (DLT).

Stratum 2 (leukemia): Patients receive dasatinib as in stratum 1. Cohorts of 3-12 patients receive escalating or de-escalating doses of dasatinib. The MTD is defined as the dose preceding that at which 7 of 12 patients experience DLT.

After completing study treatment, patients are followed for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Malignant extracranial solid tumor

    * Recurrent or refractory disease
    * Known bone marrow metastases* allowed
  * Imatinib mesylate-resistant Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia (ALL), defined as M3 bone marrow in a patient who previously received imatinib mesylate-containing treatment regimen
  * Imatinib mesylate-resistant Ph+ chronic myelogenous leukemia (CML), as defined by any of the following:

    * Increasing WBC or platelet count while on imatinib mesylate therapy
    * Lack of any cytogenetic response after an adequate duration of imatinib mesylate therapy, as defined by 1 of the following:

      * Failed to achieve a complete hematologic response after completion of 3 months of imatinib mesylate treatment
      * Failed to achieve a partial or complete cytogenetic response (i.e., ≤ 35% Ph+ cells) after 6 months of imatinib mesylate treatment
    * Appearance of accelerated or blastic feature while on imatinib mesylate therapy
    * Reappearance of Ph+ clones after an initial complete cytogenetic response to imatinib mesylate
    * More than 30% increase in Ph+ cells in peripheral blood or bone marrow cytogenetics while on imatinib mesylate therapy
    * Imatinib mesylate intolerance, as defined by development of adverse effects requiring discontinuation of imatinib mesylate therapy
* Measurable disease (for patients with CML or ALL)

  * Determined by hematologic, cytogenetic, and molecular studies for CML
  * Determined by bone marrow blast percentage for ALL
* Measurable or evaluable disease (for patients with solid tumors)
* No known curative therapy or survival-prolonging therapy with an acceptable quality of life
* No CNS solid tumors

  * CNS-positive leukemia allowed
* Karnofsky performance status (PS) ≥ 50% (for patients > 10 years of age)
* Lansky PS ≥ 50% (for patients ≤ 10 years of age)
* No evidence of graft-vs-host disease
* Solid tumors:

  * Absolute neutrophil count ≥ 1,000/mm^3 (750/mm^3 if bone marrow infiltration)
  * Platelet count ≥ 100,000/mm^3 (transfusion independent) (50,000/mm^3 if bone marrow infiltration)
  * Hemoglobin ≥ 8.0 g/dL (red blood cell [RBC] transfusions allowed)
* ALL/CML:

  * Platelet count ≥ 20,000/mm^3 (platelet transfusions allowed)
  * Hemoglobin ≥ 8.0 g/dL (RBC transfusions allowed)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine based on age, as follows:

  * No greater than 0.6 mg/dL (1-23 months of age)
  * No greater than 0.8 mg/dL (2- 5 years of age)
  * No greater than 1.0 mg/dL (6-9 years of age)
  * No greater than 1.2 mg/dL (10-12 years of age)
  * No greater than 1.4 mg/dL (13 years of age and over [female])
  * No greater than 1.5 mg/dL (13-15 years of age [male])
  * No greater than 1.7 mg/dL (16 years of age and over [male])
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 110 U/L
* Albumin ≥ 2 g/dL
* Normal 12-lead EKG with corrected QTc < 450 msec AND meets 1 of the following criteria:

  * Shortening fraction normal
  * Ejection fraction normal
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94% if there is a clinical indication for determination
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No swallowing dysfunction that would prevent taking an oral or liquid medication
* See Disease Characteristics
* Recovered from prior chemotherapy, immunotherapy, or radiotherapy
* No myelosuppressive chemotherapy within the past 3 weeks (6 weeks for nitrosoureas)
* At least 7 days since prior growth factors
* At least 14 days since prior pegfilgrastim
* At least 7 days since prior biologic agents
* At least 2 weeks since prior local small-port palliative radiotherapy
* At least 3 months since prior total-body irradiation, craniospinal radiation, or radiation to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiation
* At least 3 months since prior stem cell transplantation
* Hydroxyurea cytoreduction for Ph+ leukemia allowed provided it is discontinued 24 hours before first dose of dasatinib
* Prior intrathecal (IT) therapy allowed (for patients with CNS-positive leukemia)
* Concurrent IT therapy comprising hydrocortisone, cytarabine, methotrexate, or cytarabine (liposomal) allowed (for patients with CNS-positive leukemia)
* No other concurrent investigational drugs
* No other concurrent anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No concurrent enzyme-inducing anticonvulsants, including any of the following:

  * Phenytoin
  * Phenobarbital
  * Carbamazepine
  * Felbamate
  * Primdone
  * Oxcarbazepine
* No concurrent antithrombotic or antiplatelet agents, including any of the following:

  * Warfarin
  * Heparin
  * Low-molecular weight heparin
  * Aspirin
  * Ibuprofen
  * Other nonsteroidal anti-inflammatory drugs
* No concurrent CYP3A4 inhibitors, including itraconazole, ketoconazole, and voriconazole
* No concurrent highly active antiretroviral treatment for HIV-positive patients

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2006-03; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the maximum dose at which fewer than 1/3 patients experience dose-limiting toxicities (DLT) graded according to CTCAE | 28 days
Time to disease progression | Interval from enrollment to disease progression, death, occurrence of a second malignant neoplasm or last patient contact, assessed up to 1 month
  Will be estimated separately for patients on the solid tumor and on the refractory Ph+ leukemia strata with the Kaplan Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States